CLINICAL TRIAL: NCT06546813
Title: Outcomes of ICT Assistive Technology in RehabiliTAtIoN Pathways
Acronym: ATTAIN
Status: Recruiting | Type: Observational
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: Ministry of Health, Italy (Other Government)
Responsible Party: Principal Investigator, Claudia Salatino, Eng., Fondazione Don Carlo Gnocchi Onlus
Other Study IDs: ATTAIN
Record Dates: First submitted 2024-06-04; First posted 2024-08-09 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Communication Aids for Disabled; Communication Disorders; Motor Disorders; Cognitive Disorder
Keywords: ICT AT; AAC AT; AAL AT; Assistive Technology; Outcome Assessment
MeSH Terms: conditions — Communication Disorders; Motor Disorders; Cognitive Dysfunction | interventions — Weights and Measures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Fifty patients in need of ICT prosthetic interventions: Persons with communication, mobility or cognitive disability
  Interventions: Other: scales and questionnaire administration

INTERVENTIONS:
Other: scales and questionnaire administration — evaluation of the quality of prosthetic intervention, verification of the adequacy of assistive devices, and outcomes measurement

SUMMARY:
The study aims to improve the quality of prosthetic intervention and verify the adequacy of assistive devices, and measurement outcomes. Fifty patients in need of prosthetic interventions for Augmentative Alternative Communication, computer accessibility, and environmental control will be recruited within the DAT Unit of the Fondazione Don Carlo Gnocchi "IRCCS S.Maria Nascente" in Milan. At baseline (T0) a physician and a psychologist will perform a clinical evaluation and the AT outcome assessment. The participants will be contacted for the follow-up phase (T1) 3 to 6 months after having received the assistive solution. At T1 clinicians will readminister the AT outcome assessment. In order to make the assessment accessible to all participants, these tests and questionnaires will be administered on Windows PCs, using Grid3 software, or on a specifically created accessible web page.

DETAILED DESCRIPTION:
Fifty patients in need of prosthetic interventions for Augmentative Alternative Communication (AAC), computer accessibility, and environmental control (for example, communicators, facilitated keyboards, mouse emulators, eye pointers, accessibility software, and remote controls for home control) will be recruited within the DAT Unit of the Fondazione Don Carlo Gnocchi ONLUS "IRCCS Santa Maria Nascente" in Milan. At baseline (T0) a physician will administer the Barthel Index 20 the Modified Cumulative Illness Rating Scale (CIRS), the ICF Generic Core Set-7, the ICF-core set for profiling communicative competence for AAC AT assessments or the ICF-Vocational Rehabilitation Brief Core Set integrated with some items of the Comprehensive one for ICT AT. A psychologist will assess patients' cognitive status using the Oxford Cognitive Screening (OCS), the CPM-Coloured Progressive Matrices, the Palm and Pyramid Trees Test - short version, the Aachener Aphasie Test (AAT) subtest on written and oral comprehension of words and sentences, the Multiple Features Targets Cancellation (MFTC). In order to make the cognitive assessment accessible to all participants, these tests will be administered on Windows PCs, using The Grid3 software, or on a specifically created accessible web page. According to the clinical and cognitive assessment, the health practitioner will decide whether to administer the assessment protocol to the patient or to the closest relative. The AT assessment protocol includes at baseline: the EQ-5D-5L questionnaire for quality of life and the Individual Prioritised Problems Assessment (IPPA) to assess the importance and severity of the problems the participants expect to improve with the AT use. The DAT multidisciplinary team will conduct the AT assessment and the most appropriate assistive solution will be identified and prescribed or suggested. The assistive devices received will be classified according to the international standard ISO 9999:2016 and the Ministry of Health Prosthetics and Assistive Products List (DPCM 12/01/2017). The participants will be contacted for the follow-up phase (T1) 3 to 6 months after having received the assistive solution. At T1 clinicians will administer the IPPA questionnaire, the ICF Core Sets, the EQ-5D-5L questionnaire, and the Quebec User Evaluation of Satisfaction with Assistive Technology Questionnaire (QUEST). Quantitative data will be summarized by appropriate descriptive statistics (mean, standard deviation, median, and ranges). Qualitative data will be summarized in contingency tables.

ELIGIBILITY:
consecutive enrollment of subjects falling within

Inclusion Criteria:

* patients in need of prosthetic interventions for Augmentative Alternative Communication, computer accessibility, and environmental control
* patients who agree to participate in the study

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with mobility, communication or cognitive disability
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
QUEST-Quebec User Evaluation of Satisfaction with Assistive Technology Questionnaire | T1 (6 months)
  The "Questionnaire de Satisfaction des Usagers des Services en Travailleur Autonome" (QUEST) evaluates user satisfaction with home care and assistive technology services. It assesses:
  1. Overall Satisfaction: How well the service met expectations.
  2. Quality of Services: Perception of service quality, including provider competence and professionalism.
  3. Effectiveness: Impact on quality of life and independence.
  4. Accessibility: Ease of accessing services, considering geography, waiting times, and cost.
  5. Adequacy: How well the service met individual needs and preferences.
  6. Support and Training: Quality of support and training for using the service or technology.
  Users answer specific questions on a rating scale, helping to identify areas for improvement and optimize service quality.
IPPA-Individual Prioritised Problems Assessment | T0, T1 (3-6 months)
  Perceived effectiveness of prescribed AT
EQ-5D-5L (EuroQol - 5 Dimensions - 5 Levels) | T0, T1 (3-6 months)
  The EQ-5D-5L(EuroQol - 5 Dimensions - 5 Levels) measures health-related quality of life across five dimensions: Mobility, Self-care, Usual activities, Pain/discomfort, and Anxiety/depression. Each dimension has five severity levels ranging from "No problems" to "Extreme problems." Respondents choose a level for each dimension, resulting in a health profile of five numbers. Additionally, the scale includes a Visual Analog Scale (VAS) where overall health is rated from 0 (worst imaginable) to 100 (best imaginable). The profile can be converted into a single utility score, ranging from about -0.281 (worse than death) to 1 (perfect health). Higher scores indicate better health outcomes.

SECONDARY OUTCOMES:
Barthel Index (BI) 20 | T0, T1 (3-6 months)
  The Barthel Index (BI) - 20-point version assesses basic daily living activities to measure a patient's independence. It scores 10 activities (e.g., feeding, bathing, dressing) from 0 to 2 points each, where 0 is total dependence, 1 is partial assistance needed, and 2 is complete independence. Scores are summed to determine the level of dependence: 0-4 (total dependence), 5-9 (severe), 10-14 (moderate), 15-19 (slight), and 20 (complete independence). The index is used by healthcare professionals or caregivers through a structured questionnaire or checklist to evaluate disability, plan discharge, and monitor rehabilitation progress.
CIRS-Modified Cumulative Illness Rating Scale (CIRS-CIRS) | T0, T1 (3-6 months)
  Health condition:
  A low total score indicates good overall health with few or no significant chronic problems.
  A high total score indicates numerous severe chronic conditions, suggesting a high degree of comorbidity and a need for intensive medical intervention.
ICF (International Classification of Functioning) core-sets | T0, T1 (3-6 months)
  Classification of functioning, disability and health

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Salatino, Principal Investigator — IRCCS Fondazione Don Carlo Gnocchi ONLUS
Locations (1):
- IRCCS Fondazione Don Carlo Gnocchi ONLUS, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Borgnis F, Desideri L, Converti RM, Salatino C. Available Assistive Technology Outcome Measures: Systematic Review. JMIR Rehabil Assist Technol. 2023 Nov 15;10:e51124. doi: 10.2196/51124. PMID 37782310
- [Background] Salatino C, Andrich R, Converti RM, Saruggia M. An observational study of powered wheelchair provision in Italy. Assist Technol. 2016 Spring;28(1):41-52. doi: 10.1080/10400435.2015.1074631. PMID 26479206
- [Background] Caronni A, Ramella M, Arcuri P, Salatino C, Pigini L, Saruggia M, Folini C, Scarano S, Converti RM. The Rasch Analysis Shows Poor Construct Validity and Low Reliability of the Quebec User Evaluation of Satisfaction with Assistive Technology 2.0 (QUEST 2.0) Questionnaire. Int J Environ Res Public Health. 2023 Jan 6;20(2):1036. doi: 10.3390/ijerph20021036. PMID 36673791